CLINICAL TRIAL: NCT00110461
Title: A Phase III Trial to Test the Safety and Efficacy of Two Doses of Aripiprazole in Child and Adolescent Patients With Bipolar I Disorder, Manic or Mixed Episode With or Without Psychotic Features
Brief Title: Aripiprazole in Children and Adolescents With Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Arifulla Khan, MD, Northwest Clinical Research Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 31-03-240
Record Dates: First submitted 2005-05-09; First posted 2005-05-10 (Estimated); Results first posted 2012-05-21 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-04

CONDITIONS: Bipolar Disorder
Keywords: Aripiprazole; Bipolar I Disorder, Manic or Mixed Episode with or without Psychotic Features
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Active Comparator): Aripiprazole 10 mg tablet
  Interventions: Drug: Aripiprazole
- 2 (Active Comparator): Aripiprazole 30 mg tablet
  Interventions: Drug: Aripiprazole
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Aripiprazole — Treatment Arm 1 (10 mg treatment arm): Aripiprazole 2 mg QD for 2 days, aripiprazole 5 mg QD for 2 days, and aripiprazole 10 mg QD as the target dose starting on Day 5. Subjects remained on the 10 mg dose for the remainder of the treatment period Subjects reached their target dose through a forced titration schedule and proceeded with treatment at their target dose until Week 4. If the subject reached Week 4, he or she continued into the Extension Phase, a 6-month double-blind treatment period, beginning at the same dose taken at the end of the Acute Phase.
  Arms: 1
Drug: Aripiprazole — Treatment Arm 2 (30 mg treatment arm): Aripiprazole 2 mg QD for 2 days, aripiprazole 5 mg QD for 2 days, aripiprazole 10 mg QD for 2 days, aripiprazole 15 mg QD for 2 days, aripiprazole 20 mg QD for 2 days, aripiprazole 25 mg QD for 2 days, and aripiprazole 30 mg QD as the target dose starting on Day 13. Subjects remained on the 30 mg dose for the remainder of the treatment period. Subjects reached their target dose through a forced titration schedule and proceeded with treatment at their target dose until Week 4. If the subject reached Week 4, he or she continued into the Extension Phase, a 6-month double-blind treatment period, beginning at the same dose taken at the end of the Acute Phase.
  Arms: 2
Drug: placebo — Placebo tablet
  Arms: 3

SUMMARY:
The purpose of this trial is to test the safety and efficacy of two doses of aripiprazole in child and adolescent patients with bipolar I disorder, manic or mixed episode with or without psychotic features.

ELIGIBILITY:
Inclusion Criteria:

* Child and adolescent patients with bipolar I disorder, manic or mixed episode with or without psychotic features

Exclusion Criteria:

* Patients with certain other psychological disorders
* Patients with a co-morbid serious, uncontrolled systemic illness
* Patients with significant risk of committing suicide

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 296 (Actual)
Dates: Start 2005-03; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaretta Nyilas, MD, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (53):
- United States (53):
  - Local Institution, Scottsdale, Arizona
  - Local Institution, Little Rock, Arkansas
  - Local Institution, National City, California
  - Local Institution, Orange, California
  - Local Institution, Pasadena, California
  - Local Institution, Sacramento, California
  - Local Institution, San Diego, California
  - Local Institution, Stanford, California
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, Altamonte Springs, Florida
  - Local Institution, Hialeah, Florida
  - Local Institution, Jacksonville, Florida
  - Local Institution, Miami, Florida
  - Local Institution, North Miami, Florida
  - Local Institution, Tampa, Florida
  - Local Institution, Atlanta, Georgia
  - Local Institution, Smyrna, Georgia
  - Local Institution, Boise, Idaho
  - Local Institution, Chicago, Illinois
  - Local Institution, Libertyville, Illinois
  - Local Institution, Indianapolis, Indiana
  - Local Institution, Kansas City, Kansas
  - Local Institution, Newton, Kansas
  - Local Institution, Lexington, Kentucky
  - Local Institution, Baton Rouge, Louisiana
  - Local Institution, Lake Charles, Louisiana
  - Local Institution, Shreveport, Louisiana
  - Local Institution, Cambridge, Massachusetts
  - Local Institution, Medford, Massachusetts
  - Local Institution, Clinton Township, Michigan
  - Local Institution, Rochester Hills, Michigan
  - Local Institution, Kansas City, Missouri
  - Local Institution, St Louis, Missouri
  - Local Institution, Las Vegas, Nevada
  - Local Institution, Elmsford, New York
  - Local Institution, New York, New York
  - Local Institution, Rochester, New York
  - Local Institution, Stony Brook, New York
  - Local Institution, Cincinnati, Ohio
  - Local Institution, Cleveland, Ohio
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Charleston, South Carolina
  - Local Institution, Memphis, Tennessee
  - Local Institution, Bellaire, Texas
  - Local Institution, Fort Worth, Texas
  - Local Institution, Houston, Texas
  - Local Institution, San Antonio, Texas
  - Local Institution, Herndon, Virginia
  - Local Institution, Richmond, Virginia
  - Local Institution, Kirkland, Washington
  - Local Institution, Spokane, Washington
  - Local Institution, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Youngstrom E, Zhao J, Mankoski R, Forbes RA, Marcus RM, Carson W, McQuade R, Findling RL. Clinical significance of treatment effects with aripiprazole versus placebo in a study of manic or mixed episodes associated with pediatric bipolar I disorder. J Child Adolesc Psychopharmacol. 2013 Mar;23(2):72-9. doi: 10.1089/cap.2012.0024. Epub 2013 Mar 12. PMID 23480324
- [Derived] Findling RL, Correll CU, Nyilas M, Forbes RA, McQuade RD, Jin N, Ivanova S, Mankoski R, Carson WH, Carlson GA. Aripiprazole for the treatment of pediatric bipolar I disorder: a 30-week, randomized, placebo-controlled study. Bipolar Disord. 2013 Mar;15(2):138-49. doi: 10.1111/bdi.12042. PMID 23437959
- [Derived] Mankoski R, Zhao J, Carson WH, Mathew SJ, Forbes RA. Young mania rating scale line item analysis in pediatric subjects with bipolar I disorder treated with aripiprazole in a short-term, double-blind, randomized study. J Child Adolesc Psychopharmacol. 2011 Aug;21(4):359-64. doi: 10.1089/cap.2010.0100. Epub 2011 Aug 8. PMID 21823911
- [Derived] Findling RL, Nyilas M, Forbes RA, McQuade RD, Jin N, Iwamoto T, Ivanova S, Carson WH, Chang K. Acute treatment of pediatric bipolar I disorder, manic or mixed episode, with aripiprazole: a randomized, double-blind, placebo-controlled study. J Clin Psychiatry. 2009 Oct;70(10):1441-51. doi: 10.4088/JCP.09m05164yel. PMID 19906348

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 59 centers in the United States between March 2005 and February 2007. A total of 413 subjects were screened for enrollment, with 296 subjects assigned to double-blind treatment.
Pre-assignment Details: Participants were screened over a 28-day period.
Groups:
- Aripiprazole 10 mg/Day: Dose was titrated to a target dose of 10 mg/day as follows: Starting dose 2 mg/day, increased to 5 mg/day on Day 3, 10 mg/day on Day 5. One dose reduction to 5 mg/day was allowed in the extension phase. Following a dose reduction, the dose could be up titrated to 10 mg/day if needed.
- Aripiprazole 30 mg/Day: Dose was titrated to a target dose of 30 mg/day as follows: Starting dose 2 mg/day, increased to 5 mg/day on Day 3, 10 mg/day on Day 5, 15 mg/day on Day 7, 20 mg/day on Day 9, 25 mg/day on Day 11, and 30 mg/day on Day 13. One dose reduction to 15 mg/day was allowed in the extension phase. Following a dose reduction, the dose could be up titrated to 20 mg/day if needed.
- Placebo: Participants were given a single pill administered once daily.
Period: 30-Week, Double-blind Treatment Phase
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Started | 98 | 99 | 99
Completed | 34 | 22 | 12
Not Completed | 64 | 77 | 87
Period: Acute Phase
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Started | 98 | 99 | 99
Completed | 84 | 77 | 76
Not Completed | 14 | 22 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo | Total
Number analyzed (Participants) | 98 | 99 | 99 | 296
Age Continuous [Mean (Standard Deviation); unit: years] | 13.70 (2.17) | 13.31 (2.32) | 13.28 (2.12) | 13.43 (2.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 48 | 43 | 137
  Male | 52 | 51 | 56 | 159
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 10 | 15 | 31
  Not Hispanic or Latino | 92 | 89 | 84 | 265
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 2
  Black or African American | 24 | 18 | 23 | 65
  White | 65 | 68 | 60 | 193
  More than one race | 2 | 2 | 2 | 6
  Unknown or Not Reported | 5 | 11 | 14 | 30
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 161.05 (12.45) | 158.37 (12.21) | 158.69 (11.63) | 159.36 (12.12)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 63.76 (20.11) | 60.49 (21.50) | 60.48 (17.31) | 61.57 (19.71)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.15 (5.37) | 23.66 (6.70) | 23.68 (4.98) | 23.83 (5.72)
Young Mania Rating Scale Score (Y-MRS) [Mean (Standard Deviation); unit: points] — The Y-MRS consists of 11 items assessing the core symptoms of mania. Each item has 5 defined grades of severity. Minimum score on the scale is 0 (absent or normal); maximum score on the scale is 60 (worse outcome or more severe symptoms).
  points | 29.8 (6.5) | 29.5 (6.3) | 30.7 (6.8) | 30.0 (6.5)
Children's Depression Rating Scale - Revised (CDRS-R) Suicidal Ideation Score [Mean (Standard Deviation); unit: points] — The CDRS-R is used to diagnose depression and monitor treatment response. The interviewer rates 17 symptom areas (including those that sever as DSM-IV criteria for diagnosis of depression), among them suicidal ideation. Most of the 17 symptom areas are rated on a 7-point scale. The Suicide Ideation Score is rated on a 7-point scale, where the minimum score on the scale is 1 (better outcome) and the maximum score is 7 (worse outcome).
  points | 1.1 (0.4) | 1.1 (0.5) | 1.2 (0.5) | 1.2 (0.5)
Treatment given for previous episodes [Number; unit: participants]
  Yes | 57 | 50 | 63 | 170
  No | 41 | 49 | 36 | 126

OUTCOME MEASURES:

1. Primary Outcome: Change in Young Mania Rating Scale (Y-MRS) Total Score at Week 4
Description: Change from Baseline to Week 4 in Y-MRS total score, using the last observation carried forward.
  Assessments performed at baseline and weekly through the acute phase (Week 4). (Also performed at Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through the continuation phase.)
  The Y-MRS consists of 11 items assessing the core symptoms of mania. Each item has 5 grades of severity. Minimum score on the scale is 0 (absent or normal). Maximum score on the scale is 60 (worse outcome or more severe symptoms).
Time Frame: Baseline and Week 4
Population: Since the primary efficacy endpoint is change from baseline in Y-MRS total score, only randomized subjects who had both baseline and at least one post-baseline were included in the primary efficacy analysis. Therefore, number of randomized subjects be different number subjects included in the efficacy analysis.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 96 | 99 | 92
points | -14.04 (9.33) [-8.49 to -3.50] | -16.16 (9.18) [-10.7 to -5.77] | -8.67 (9.17)
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; The change scores were analyzed by using ANCOVA model with treatment as a factor and baseline Y-MRS total score as a covariate. For comparing YMRS-Total score in treatment groups at baseline, only treatment was included in the ANOVA model with baseline values as the dependent variable. The LS means obtained from a type III analysis using SAS were used for the treatment comparisons. Two-tailed student's t-tests were used to test differences between the LS means within the ANCOVA or ANOVA model; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -5.99, 95% CI 2-sided [-8.49 to -3.5]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Median Difference (Final Values) = -8.26, 95% CI 2-sided [-10.7 to -5.77]

2. Secondary Outcome: Change in Young Mania Rating Scale (Y-MRS) Total Score at Week 30
Description: Change from baseline to Week 30 in Y-MRS total score, using the last observation carried forward.
  Assessments performed at baseline and weekly through the acute phase (Week 4) and at Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through continuation phase.
  The Y-MRS consists of 11 items assessing the core symptoms of mania. Each item has 5 grades of severity. Minimum score on the scale is 0 (absent or normal). Maximum score on the scale is 60 (worse outcome or more severe symptoms).
Time Frame: Baseline and Week 30
Population: Since the endpoint is change from baseline in Y-MRS total score, only randomized subjects who had both baseline and at least one post-baseline were included in the primary efficacy analysis. Therefore, number of randomized subjects could be different number subjects included in the efficacy analysis.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 96 | 99 | 94
points | -13.91 (10.83) | -14.6 (10.35) | -8.69 (9.88)
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; Analyses were performed by fitting an ANCOVA model with treatment as factor and baseline score as covariate. Two pair-wise comparisons, aripiprazole 10 mg target dose versus placebo and aripiprazole 30 mg target dose versus placebo, were performed within the ANCOVA or ANOVA model; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Median Difference (Final Values) = -5.89, 95% CI 2-sided [-8.7 to -3.08]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Median Difference (Final Values) = 11.51, 95% CI 2-sided [7.99 to 15.03]

3. Secondary Outcome: Change in Children's Global Assessment Scale (CGAS) Total Score at Week 4
Description: Change from baseline to Week 4 in CGAS total score, using the last observation carried forward. Assessments performed at baseline and weekly through the acute phase (Week 4). (Also performed at Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through continuation phase.)
  The CGAS is a 100-point scale measuring psychological, social, and school functioning for children aged 6 to 17 years. Minimum scores ranged from 1-10, representing the need for constant supervision (worse outcome) to maximum scores of 91-100, representing superior functioning (better outcome).
Time Frame: Baseline and Week 4
Population: Since the endpoint is change from baseline, only randomized subjects who had both baseline and at least one post-baseline were included in the efficacy analysis. Therefore, number of randomized subjects could be a different number subjects included in the efficacy analysis.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 96 | 99 | 92
points | 14.97 (14.94) | 16.96 (13.4) | 6.21 (9.15)
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Median Difference (Final Values) = 9.30, 95% CI 2-sided [5.77 to 12.84]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Median Difference (Final Values) = 11.51, 95% CI 2-sided [7.99 to 15.03]

4. Secondary Outcome: Change in Clinical Global Impressions Scale-Bipolar Version (CGI-BP) Severity Mania Score at Week 4
Description: Change from baseline to Week 4 in CGI-BP mania score, using the last observation carried forward.
  Assessments performed at baseline and weekly through the acute phase (Week 4). (Also performed at Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through continuation phase.)
  The CGI-BP scale refers to the global impression of the subject with respect to bipolar disorder. The scale rates the subject's severity of illness for mania, depression, and overall bipolar illness from 1 (least severe) to 7 (most severe).
Time Frame: Baseline and Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 96 | 99 | 92
points | -1.6 (1.3) | -2.02 (1.29) | -0.89 (1.11)
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -0.81, 95% CI 2-sided [-1.15 to -0.48]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -1.26, 95% CI [-1.59 to -0.93]

5. Secondary Outcome: Change in Children's Depression Rating Scale-Revised (CDRS-R) Total Score at Week 4
Description: Change from baseline to Week 4 in CDRS-R score, using last observation carried forward. Assessments performed at baseline and weekly through the acute phase (Week 4). (Also performed at Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through continuation phase.) The CDRS-R is used to diagnose depression and monitor treatment response. The interviewer rates 17 symptom areas (including those that sever as DSM-IV criteria for diagnosis of depression), among them suicidal ideation. Minimum score on the scale is 17 (better outcome). Maximum score on the scale is 113 (worse outcome or more severe symptoms).
Time Frame: Baseline and Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 91 | 94 | 85
points | -7.65 (11.05) | -5.97 (10.88) | -4.66 (9.1)
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0767, t-test, 2 sided; Mean Difference (Final Values) = -2.28, 95% CI 2-sided [-4.81 to 0.25]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.3515, t-test, 2 sided; Mean Difference (Final Values) = -1.19, 95% CI 2-sided [-3.69 to 1.32]

6. Secondary Outcome: Change in General Behavior Inventory Scale (GBI) Total Parent/Guardian Version Mania Score at Week 4
Description: Change from baseline to Week 4 in GBI Total Parent/Guardian Version Mania score, using LOCF. Assessments performed baseline and weekly through acute phase (Week 4). (Also at Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through continuation phase.) GBI is self-report inventory with 73 items focused on mood-related behaviors including depressive, hypomanic, and biphasic symptoms. One 20-item subscale was completed by parent/guardian. Symptoms rated on a 4-point Likert scale from 0 (never or hardly ever) to 3 (often or almost constantly). Minimum score 0=better outcome, maximum score 60=worse outcome.
Time Frame: Baseline and Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 96 | 96 | 91
points | -9.66 (9.14) | -9.1 (7.91) | -4.63 (8.97)
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -5.88, 95% CI 2-sided [-8.02 to -3.73]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -5.46, 95% CI 2-sided [-7.40 to -3.32]

7. Secondary Outcome: Change in Attention Deficit Hyperactivity Disorders Rating Scale (ADHD-RS-IV) Total Score at Week 4
Description: Change from baseline to Week 4 in ADHD-RS-IV Total score, using last observation carried forward. Assessments performed at baseline and weekly through acute phase (Week 4). (Also performed at Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through continuation phase.) ADHD-RS-IV is an instrument for diagnosing ADHD in children/adolescents and for assessing treatment response. The scale contains 18 items linked directly to DSM-IV diagnostic criteria for ADHD. Parent questionnaire on home behaviors (Eng.) used in this study. Minimum score of 0 is a better outcome, maximum score of 54 is a worse outcome.
Time Frame: Baseline and Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 95 | 97 | 90
points | -12.03 (13.09) | -11.61 (14.06) | -4.57 (9.88)
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; Analyses were performed by fitting an ANCOVA model with treatment as factor, and baseline score as covariate. Two pair-wise comparisons, aripiprazole 10 mg target dose versus placebo and aripiprazole 30 mg target dose versus placebo, were performed within the ANCOVA or ANOVA model; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -8.86, 95% CI 2-sided [-12.3 to -5.43]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -8.23, 95% CI 2-sided [-11.6 to -4.83]

8. Secondary Outcome: Change in Children's Global Assessment (CGAS) Total Score at Week 30
Description: Change from baseline to Week 30 in CGAS total score, using the last observation carried forward.
  Assessments performed at baseline and weekly through the acute phase (Week 4) and at Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through continuation phase.
  The CGAS is a 100-point scale measuring psychological, social, and school functioning for children aged 6 to 17 years. Minimum scores ranged from 1-10, representing the need for constant supervision (worse outcome) to maximum scores of 91-100, representing superior functioning (better outcome).
Time Frame: Baseline and Week 30
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 96 | 99 | 94
points | 15.81 (18.81) | 16.28 (14.73) | 7.45 (11.59)
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 9.23, 95% CI 2-sided [5.07 to 13.93]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Median Difference (Final Values) = 10, 95% CI 2-sided [5.87 to 14.14]

9. Secondary Outcome: Change in Clinical Global Impressions Scale-Bipolar Version (CGI-BP) Severity Mania Score at Week 30
Description: Change from baseline to Week 30 in CGI-BP mania score, using the last observation carried forward.
  Assessments performed at baseline and weekly through the acute phase (Week 4) and at Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through continuation phase.
  The CGI-BP scale refers to the global impression of the subject with respect to bipolar disorder. The scale rates the subject's severity of illness for mania, depression, and overall bipolar illness from 1 (least severe) to 7 (most severe).
Time Frame: Baseline and Week 30
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 96 | 99 | 94
points | -1.63 (1.43) | -1.93 (1.4) | -1.03 (1.32)
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0003, t-test, 2 sided; Median Difference (Final Values) = -0.70, 95% CI 2-sided [-1.08 to -0.33]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Median Difference (Final Values) = -1.04, 95% CI 2-sided [-1.41 to -0.66]

10. Secondary Outcome: Change in Clinical Global Impressions Scale-Bipolar Version (CGI-BP) Severity Depression Score at Week 4
Description: Change from baseline to Week 4 in CGI-BP severity depression score, using the last observation carried forward.
  Assessments performed at baseline and weekly through the acute phase (Week 4. (Also performed at Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through continuation phase.)
  The CGI-BP scale refers to the global impression of the subject with respect to bipolar disorder. The scale rates the subject's severity of illness for mania, depression, and overall bipolar illness from 1 (least severe) to 7 (most severe).
Time Frame: Baseline and Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 96 | 99 | 92
points | -0.86 (1.37) | -0.9 (1.32) | -0.57 (1.21)
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0878, t-test, 2 sided; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.54 to 0.04]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0752, t-test, 2 sided; Median Difference (Final Values) = -0.26, 95% CI 2-sided [-0.55 to 0.03]

11. Secondary Outcome: Change in Clinical Global Impressions Scale-Bipolar Version (CGI-BP) Severity Depression Score at Week 30
Description: Change from baseline to Week 30 in CGI-BP severity depression score, using the last observation carried forward.
  Assessments performed at baseline and weekly through the acute phase (Week 4) and at Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through continuation phase.
  The CGI-BP scale refers to the global impression of the subject with respect to bipolar disorder. The scale rates the subject's severity of illness for mania, depression, and overall bipolar illness from 1 (least severe) to 7 (most severe).
Time Frame: Baseline and Week 30
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 96 | 99 | 94
points | -0.71 (1.44) | -0.94 (1.38) | -0.47 (1.45)
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2553, t-test, 2 sided; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.51 to 0.13]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0166, t-test, 2 sided; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-0.71 to -0.07]

12. Secondary Outcome: Change in Clinical Global Impressions Scale-Bipolar Version (CGI-BP) Severity Overall Illness Score at Week 4
Description: Change from baseline to Week 4 in CGI-BP severity overall illness score, using the last observation carried forward.
  Assessments performed at baseline and weekly through the acute phase (Week 4). (Also performed and at Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through continuation phase.)
  The CGI-BP scale refers to the global impression of the subject with respect to bipolar disorder. The scale rates the subject's severity of illness for mania, depression, and overall bipolar illness from 1 (least severe) to 7 (most severe).
Time Frame: Baseline and Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 96 | 99 | 92
points | -1.6 (1.33) | -1.91 (1.21) | -0.84 (1.02)
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-1.16 to -0.51]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Median Difference (Final Values) = -1.18, 95% CI 2-sided [-1.51 to -0.86]

13. Secondary Outcome: Change in Clinical Global Impressions Scale-Bipolar Version (CGI-BP) Severity Overall Illness Score at Week 30
Description: Change from baseline to Week 30 in CGI-BP severity overall illness score, using the last observation carried forward.
  Assessments performed at baseline and weekly through the acute phase (Week 4) and at Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through continuation phase.
  The CGI-BP scale refers to the global impression of the subject with respect to bipolar disorder. The scale rates the subject's severity of illness for mania, depression, and overall bipolar illness from 1 (least severe) to 7 (most severe).
Time Frame: Baseline and Week 30
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 96 | 99 | 94
points | -1.59 (1.45) | -1.75 (1.34) | -0.91 (1.24)
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -0.76, 95% CI 2-sided [-1.13 to -0.40]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -0.97, 95% CI 2-sided [-1.33 to -0.60]

14. Secondary Outcome: Change in Children's Depression Rating Scale-Revised (CDRS-R) Total Score at Week 30
Description: Change from baseline to Week 30 in CDRS-R score, using the last observation carried forward. Assessments performed at baseline and weekly through the acute phase (Week 4) and at Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through continuation phase. The CDRS-R is used to diagnose depression and monitor treatment response. The interviewer rates 17 symptom areas (including those that sever as DSM-IV criteria for diagnosis of depression), among them suicidal ideation. Minimum score on the scale is 17 (better outcome). Maximum score on the scale is 113 (worse outcome or more severe symptoms).
Time Frame: Baseline and Week 30
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 91 | 94 | 86
points | -6.47 (11.74) | -4.39 (10.61) | -3.81 (10.91)
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.1729, t-test, 2 sided; Median Difference (Final Values) = -1.92, 95% CI 2-sided [-4.69 to 0.85]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.75586, t-test, 2 sided; Median Difference (Final Values) = -0.43, 95% CI 2-sided [-3.17 to 2.31]

15. Secondary Outcome: Change in General Behavior Inventory Scale (GBI) Total Parent/Guardian Version Mania Score at Week 30
Description: Change from baseline to Week 30 in GBI Total Parent/Guardian Version Mania score, using LOCF. Assessments performed at baseline and weekly through acute phase(Week 4) and Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through continuation phase. GBI is a self-report inventory with 73 items focused on mood-related behaviors including depressive, hypomanic, and biphasic symptoms. One 20-item subscale was completed by parent/guardian. Symptoms rated on a 4-point Likert scale from 0 (never or hardly ever) to 3 (often or almost constantly). Minimum score 0=better outcome, maximum score 60=worse outcome.
Time Frame: Baseline and Week 30
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 95 | 96 | 93
points | -8.76 (9.12) | -8.48 (8.44) | -5 (9.33)
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -4.76, 95% CI 2-sided [-6.90 to -2.61]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -4.64, 95% CI 2-sided [-6.78 to -2.50]

16. Secondary Outcome: Change in General Behavior Inventory Scale (GBI) Total Subject Version Mania Score at Week 4
Description: Change from baseline to Week 4 in GBI Total Subject Version Mania score, using the LOCF. Assessments performed at baseline and weekly through acute phase (Week 4). (Also performed Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through continuation phase.) GBI is a self-report inventory with 73 items focused on mood-related behaviors including depressive, hypomanic, and biphasic symptoms. One 20-item subscale completed by the subject. Symptoms rated on a 4-point Likert scale from 0 (never or hardly ever) to 3 (often or almost constantly). Minimum score 0=better outcome, maximum score 60=worse outcome.
Time Frame: Baseline and Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 96 | 96 | 91
points | -6.51 (7.49) | -6.52 (7.49) | -4.57 (7.21)
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.0468, t-test, 2 sided; Mean Difference (Final Values) = -1.85, 95% CI 2-sided [-3.67 to -0.03]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.0296, t-test, 2 sided; Mean Difference (Final Values) = -2.03, 95% CI 2-sided [-3.85 to -0.20]

17. Secondary Outcome: Change in General Behavior Inventory Scale (GBI) Total Subject Version Mania Score at Week 30
Description: Change from baseline to Week 30 in GBI Total Subject Version Mania score, using LOCF. Assessments performed at baseline and weekly through acute phase (Week 4) and Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through continuation phase. GBI is a self-report inventory with 73 items focused on mood-related behaviors including depressive, hypomanic, and biphasic symptoms. One 20-item subscale completed by the subject. Symptoms rated on a 4-point Likert scale from 0 (never or hardly ever) to 3 (often or almost constantly). Minimum score of 0=better outcome, maximum score of 60=worse outcome.
Time Frame: Baseline and Week 30
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 96 | 96 | 93
points | -6.82 (7.86) | -7.84 (7.7) | -5.23 (7.68)
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.1309, t-test, 2 sided; Mean Difference (Final Values) = -1.44, 95% CI 2-sided [-3.31 to 0.43]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.0058, t-test, 2 sided; Mean Difference (Final Values) = -2.64, 95% CI 2-sided [-4.51 to -0.77]

18. Secondary Outcome: Change in General Behavior Inventory Scale (GBI) Total Parent/Guardian Version Depression Score at Week 4
Description: Change from baseline to Week 4 in GBI Total Parent/Guardian Version Depression score, using LOCF. Assessments performed at baseline and weekly through the acute phase (Week 4); also Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through continuation phase. GBI is a self-report inventory with 73 items focused on mood-related behaviors including depressive, hypomanic, and biphasic symptoms. One 20-item subscale was completed by parent/guardian. Symptoms rated on 4-point Likert scale from 0 (never/hardly ever) to 3 (often/almost constantly). Minimum score 0=better outcome, maximum score 60=worse outcome.
Time Frame: Baseline and Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 95 | 96 | 91
points | -6.12 (8.78) | -3.71 (8.62) | -3.92 (8.82)
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.0430, t-test, 2 sided; Mean Difference (Final Values) = -2.13, 95% CI 2-sided [-4.20 to -0.07]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.7696, t-test, 2 sided; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-2.37 to 1.76]

19. Secondary Outcome: Change in General Behavior Inventory Scale (GBI) Total Parent/Guardian Version Depression Score at Week 30
Description: Change from Baseline to Week 30 in GBI Total Parent/Guardian Version Depression score, using LOCF. Assessments performed at baseline and weekly through the acute phase (Week 4); also Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through continuation phase. GBI is a self-report inventory with 73 items focused on mood-related behaviors including depressive, hypomanic, and biphasic symptoms. One 20-item subscale completed by parent/guardian. Symptoms rated on 4-point Likert scale from 0 (never/hardly ever) to 3 (often/almost constantly). Minimum score 0=better outcome, maximum score 60=worse outcome.
Time Frame: Baseline and Week 30
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 96 | 96 | 91
points | -5.17 (9.13) | -3.71 (9) | -3.03 (9.27)
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.9418, t-test, 2 sided; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-1.73 to 1.86]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.19, t-test, 2 sided; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-1.67 to 1.98]

20. Secondary Outcome: Change in General Behavior Inventory Scale (GBI) Total Subject Version Depression Score at Week 4
Description: Change from Baseline to Week 4 in GBI Total Subject Version Depression score, using LOCF. Assessments performed at baseline and weekly through the acute phase (Week 4); also at Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through continuation phase. GBI is a self-report inventory with 73 items focused on mood-related behaviors including depressive, hypomanic, and biphasic symptoms. One 20-item subscale was completed by subject. Symptoms wrated on a 4-point Likert scale from 0 (never or hardly ever) to 3 (often or almost constantly). Minimum score 0=better outcome, maximum score 60=worse outcome.
Time Frame: Baseline and Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 96 | 96 | 91
points | 0 (6.87) | -3.24 (6.96) | -3.11 (7.73)
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.9418, t-test, 2 sided; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-1.73 to 1.86]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.8377, t-test, 2 sided; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-1.61 to 1.98]

21. Secondary Outcome: Change in General Behavior Inventory Scale (GBI) Total Subject Version Depression Score at Week 30
Description: Change from baseline to Week 30 in GBI Total Subject Version Depression score, using LOCF. Assessments performed at baseline and weekly through the acute phase (Week 4); also at Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through continuation phase. GBI is a self-report inventory with 73 items focused on mood-related behaviors including depressive, hypomanic, and biphasic symptoms. One 20-item subscale completed by the subject. Symptoms rated on a 4-point Likert scale from 0 (never or hardly ever) to 3 (often or almost constantly). Minimum score 0=better outcome, maximum score 60=worse outcome.
Time Frame: Baseline and Week 30
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 96 | 96 | 93
points | -4.45 (7.62) | -4.38 (8.09) | -2.7 (8.44)
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.3969, t-test, 2 sided; Mean Difference (Final Values) = -0.82, 95% CI 2-sided [-2.71 to 1.08]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.2101, t-test, 2 sided; Mean Difference (Final Values) = -1.21, 95% CI 2-sided [-3.09 to 0.68]

22. Secondary Outcome: Change in Attention Deficit Hyperactivity Disorders Rating Scale (ADHD-RS-IV) Total Score at Week 30
Description: Change from baseline to Week 30 in ADHD-RS-IV Total score, using the LOCF.
  Assessments performed at baseline and weekly through the acute phase (Week 4) and at Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through continuation phase.
  The ADHD-RS-IV is an instrument both for diagnosing ADHD in children and adolescents and for assessing treatment response. The scale contains 18 items and is linked directly to DSM-IV diagnostic criteria for ADHD. The parent questionnaire on home behaviors (English) was used in this study. Minimum score of 0 = better outcome, maximum score of 54 = worse outcome.
Time Frame: Baseline and Week 30
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 95 | 97 | 91
points | -11.04 (19.32) | -9.76 (13.44) | -5.58 (10.9)
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -7.05, 95% CI 2-sided [-10.5 to -3.64]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.0014, t-test, 2 sided; Mean Difference (Final Values) = -5.55, 95% CI 2-sided [-8.94 to -2.16]

23. Secondary Outcome: Subject Response to Treatment at Week 4
Description: Percentage of Subjects with a 50% or higher reduction from baseline in Young Mania Rating Scale (Y-MRS) total score at Week 4.
  Assessments performed at baseline and weekly through the acute phase (Week 4). (Also performed at Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through continuation phase.)
  The Y-MRS consists of 11 items assessing the core symptoms of mania. Each item has 5 grades of severity. Minimum score on the scale is 0 (absent or normal). Maximum score on the scale is 60 (worse outcome or more severe symptoms).
Time Frame: Baseline and Week 4
Population: Since the primary efficacy endpoint is change from baseline in Y-MRS total score, only randomized subjects who had both baseline and at least one post-baseline were included in the primary efficacy analysis. Therefore, number of randomized subjects could be different number subjects included in the efficacy analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 96 | 99 | 92
percentage of participants | 44.79 | 63.64 | 26.09
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; Analyzed using a Chi-square test. Ninety five percent confidence intervals for difference in the responder rates are derived from the normal approximation to binomial; Test type: Superiority or Other; p = 0.0074, Chi-squared; Mean Difference (Final Values) = 18.70, 95% CI 2-sided [5.01 to 32.40]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p < 0.0001, Chi-squared; Mean Difference (Final Values) = 37.55, 95% CI 2-sided [23.41 to 51.68]

24. Secondary Outcome: Subject Response to Treatment at Week 30
Description: Percentage of Subjects with a 50% or higher reduction from baseline in Y-MRS total score at Week 30.
  Assessments performed at baseline and weekly through the acute phase (Week 4) and at Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through continuation phase.
  The Y-MRS consists of 11 items assessing the core symptoms of mania. Each item has 5 grades of severity. Minimum score on the scale is 0 (absent or normal). Maximum score on the scale is 60 (worse outcome or more severe symptoms).
Time Frame: Baseline and Week 30
Population: as for outcome 23
Measure: Number; unit: percentage of participants
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 96 | 99 | 94
percentage of participants | 50.00 | 55.56 | 26.60
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.0009, Chi-squared; Mean Difference (Final Values) = 23.40, 95% CI 2-sided [9.57 to 37.24]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p < 0.0001, Chi-squared; Mean Difference (Final Values) = 28.96, 95% CI 2-sided [15.05 to 42.87]

25. Secondary Outcome: Change From Previous Phase in Clinical Global Impressions Scale-Bipolar Version (CGI-BP) Severity Mania Score at Week 4
Description: Change from previous phase to Week 4 in CGI-BP mania score, using the last observation carried forward.
  Assessments performed at baseline and weekly through the acute phase (Week 4). (Also performed at Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through continuation phase.)
  The CGI-BP scale refers to the global impression of the subject with respect to bipolar disorder. The scale rates the change from the preceding phase score for mania, depression, and overall bipolar illness from 1 (very much improved) to 7 (very much worse).
Time Frame: Baseline and Week 4
Population: Since the endpoint is change from previous phase, only randomized subjects who had both previous phase and at least one next phase were included in the efficacy analysis. Therefore, number of randomized subjects could be a different number subjects included in the efficacy analysis.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 96 | 99 | 92
points | 2.4 (1.04) | 2.32 (1.25) | 3.37 (1.16)
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; Analyzed using the Cochran-Mantel-Haenszel row mean score statistic by week; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -0.97, 95% CI 2-sided [-1.29 to -0.66]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; Analyzed using the Cochran-Mantel-Haenszel row mean score statistic by week; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -1.05, 95% CI 2-sided [-1.39 to -0.70]

26. Secondary Outcome: Change From Previous Phase in Clinical Global Impressions Scale-Bipolar Version (CGI-BP) Severity Mania Score at Week 30
Description: Change from previous phase to Week 30 in CGI-BP mania score, using the last observation carried forward.
  Assessments performed at baseline and weekly through the acute phase (Week 4) and at Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through continuation phase.
  The CGI-BP scale refers to the global impression of the subject with respect to bipolar disorder. The scale rates the change from the preceding phase score for mania, depression, and overall bipolar illness from 1 (very much improved) to 7 (very much worse).
Time Frame: Baseline and Week 30
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 96 | 99 | 94
points | 2.61 (1.43) | 2.45 (1.39) | 3.26 (1.35)
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; Analyzed using the Cochran-Mantel-Haenszel row mean score statistic by week; Test type: Superiority or Other; p = 0.0020, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -0.64, 95% CI 2-sided [-1.04 to -0.24]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -0.80, 95% CI 2-sided [-1.19 to -0.41]

27. Secondary Outcome: Change From Previous Phase in Clinical Global Impressions Scale-Bipolar Version (CGI-BP) Severity Depression Score at Week 4
Description: Change from previous phase to Week 4 in CGI-BP severity depression score, using the last observation carried forward.
  Assessments performed at baseline and weekly through the acute phase (Week 4). (Also performed at Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through continuation phase.)
  The CGI-BP scale refers to the global impression of the subject with respect to bipolar disorder. The scale rates the change from the preceding phase score for mania, depression, and overall bipolar illness from 1 (very much improved) to 7 (very much worse).
Time Frame: Baseline and Week 4
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 96 | 99 | 92
points | 2.96 (1.27) | 3.06 (1.26) | 3.57 (1.19)
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; Analyzed using the Cochran-Mantel-Haenszel row mean score statistic by week; Test type: Superiority or Other; p = 0.0010, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-0.96 to -0.26]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; Analyzed using the Cochran-Mantel-Haenszel row mean score statistic by week; Test type: Superiority or Other; p = 0.0053, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-0.85 to -0.16]

28. Secondary Outcome: Change From Previous Phase in Clinical Global Impressions Scale-Bipolar Version (CGI-BP) Severity Depression Score at Week 30
Description: Change from previous phase to Week 30 in CGI-BP severity depression score, using the last observation carried forward.
  Assessments performed at baseline and weekly through the acute phase (Week 4) and at Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through continuation phase.
  The CGI-BP scale refers to the global impression of the subject with respect to bipolar disorder. The scale rates the change from the preceding phase score for mania, depression, and overall bipolar illness from 1 (very much improved) to 7 (very much worse).
Time Frame: Baseline and Week 30
Population: Since the endpoint is change from previous week, only randomized subjects who had both previous week and at least next week were included in the efficacy analysis. Therefore, number of randomized subjects could be a different number subjects included in the efficacy analysis.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 96 | 99 | 94
points | 3.3 (1.33) | 3.06 (1.14) | 3.56 (1.31)
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; Analyzed using the Cochran-Mantel-Haenszel row mean score statistic by week; Test type: Superiority or Other; p = 0.1726, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.64 to 0.11]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; Analyzed using the Cochran-Mantel-Haenszel row mean score statistic by week; Test type: Superiority or Other; p = 0.0113, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-0.89 to -0.12]

29. Secondary Outcome: Change From Previous Phase in Clinical Global Impressions Scale-Bipolar Version (CGI-BP) Severity Overall Illness Score at Week 4
Description: Change from previous phase to Week 4 in CGI-BP severity overall illness score, using the last observation carried forward.
  Assessments performed at baseline and weekly through the acute phase (Week 4). (Also performed at Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through continuation phase.)
  The CGI-BP scale refers to the global impression of the subject with respect to bipolar disorder. The scale rates the change from the preceding phase score for mania, depression, and overall bipolar illness from 1 (very much improved) to 7 (very much worse).
Time Frame: Baseline and Week 4
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 96 | 99 | 92
points | 2.48 (1.09) | 2.41 (1.2) | 3.47 (1.17)
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; Analyzed using the Cochran-Mantel-Haenszel row mean score statistic by week; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -0.99, 95% CI 2-sided [-1.31 to -0.67]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; Analyzed using the Cochran-Mantel-Haenszel row mean score statistic by week; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -1.05, 95% CI 2-sided [-1.39 to -0.72]

30. Secondary Outcome: Change From Previous Phase in Clinical Global Impressions Scale-Bipolar Version (CGI-BP) Severity Overall Illness Score at Week 30
Description: Change from previous phase to Week 30 in CGI-BP severity overall illness score, using the last observation carried forward.
  Assessments performed at baseline and weekly through the acute phase (Week 4) and at Weeks 6, 8, 10, 12, 16, 20, 24, and 30 through continuation phase.
  The CGI-BP scale refers to the global impression of the subject with respect to bipolar disorder. The scale rates the change from the preceding phase score for mania, depression, and overall bipolar illness from 1 (very much improved) to 7 (very much worse).
Time Frame: Baseline and Week 30
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Number analyzed (Participants) | 96 | 99 | 94
points | 2.75 (1.49) | 2.6 (1.38) | 3.38 (1.38)
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day vs Placebo; Analyzed using the Cochran-Mantel-Haenszel row mean score statistic by week; Test type: Superiority or Other; p = 0.0030, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -0.63, 95% CI 2-sided [-1.04 to -0.22]
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day vs Placebo; Analyzed using the Cochran-Mantel-Haenszel row mean score statistic by week; Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -0.79, 95% CI 2-sided [-1.18 to -0.40]

ADVERSE EVENTS:
Arm/Group | Aripiprazole 10 mg/Day | Aripiprazole 30 mg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 5/98 | 7/99 | 6/97
Other Adverse Events (participants affected / at risk) | 78/98 | 84/99 | 64/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole 10 mg/Day (N=98) | Aripiprazole 30 mg/Day (N=99) | Placebo (N=97)
Fatigue (General disorders) | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0 | 0
Agression (Psychiatric disorders) | 2 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 5 | 4
Bipolar I disorder (Psychiatric disorders) | 0 | 2 | 1
Libido increased (Psychiatric disorders) | 0 | 1 | 0
Mania (Psychiatric disorders) | 0 | 0 | 1
Oppositional defiant disorder (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole 10 mg/Day (N=98) | Aripiprazole 30 mg/Day (N=99) | Placebo (N=97)
Vision blurred (Eye disorders) | 10 | 8 | 1
Abdominal pain (Gastrointestinal disorders) | 9 | 5 | 3
Diarrhea (Gastrointestinal disorders) | 4 | 5 | 0
Nausea (Gastrointestinal disorders) | 13 | 14 | 5
Salivary hypersecretion (Gastrointestinal disorders) | 3 | 8 | 0
Stomach discomfort (Gastrointestinal disorders) | 2 | 6 | 2
Vomiting (Gastrointestinal disorders) | 13 | 8 | 9
Fatigue (General disorders) | 18 | 12 | 4
Nasopharyngitis (Infections and infestations) | 7 | 3 | 3
Upper respiratory tract infection (Infections and infestations) | 8 | 6 | 3
Weight increased (Investigations) | 8 | 5 | 3
Decreased appetite (Metabolism and nutrition disorders) | 7 | 4 | 3
Increased appetite (Metabolism and nutrition disorders) | 8 | 8 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 3 | 2
Akathisia (Nervous system disorders) | 9 | 13 | 2
Dizziness (Nervous system disorders) | 7 | 5 | 1
Dystonia (Nervous system disorders) | 2 | 5 | 0
Extrapyramidal disorder (Nervous system disorders) | 12 | 28 | 3
Headache (Nervous system disorders) | 20 | 23 | 18
Somnolence (Nervous system disorders) | 24 | 27 | 3
Anxiety, upper (Psychiatric disorders) | 5 | 1 | 3
Bipolar disorder (Psychiatric disorders) | 0 | 6 | 5
Insomnia (Psychiatric disorders) | 6 | 1 | 2
Dysmenorrhea (Reproductive system and breast disorders) | 5 | 0 | 2
Cough, upper (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 | 3 | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 3

LIMITATIONS AND CAVEATS:
Primary efficacy endpoint is change from baseline in Y-MRS total score. Only randomized subjects with both baseline and 1+ post-baseline were included in primary efficacy analysis so # randomized is different from # included in the efficacy analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs may not publish trial results for 18 months - 2 years after trial is completed.